CLINICAL TRIAL: NCT07138482
Title: Health Literacy and Social Determinants of Health (SDOH) in the Perioperative Setting
Brief Title: Health Literacy in the Perioperative Setting
Status: Recruiting | Type: Observational
Sponsor: Brittany Willer (Other)
Responsible Party: Sponsor-Investigator, Brittany Willer, Pediatric Anesthesiologist, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00004902
Record Dates: First submitted 2025-07-02; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Pediatric Surgery; Health Literacy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey using a questionnaire. — REDCap Survey

SUMMARY:
The purpose of this study is to determine the association of the social determinants of health with perioperative health literacy in caregivers of children presenting for surgery. Another purpose is to determine the association of caregiver health literacy with preoperative caregiver anxiety and postoperative patient pain scores.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children age 3-17 years
* Patient undergoing ambulatory dental rehabilitation, orchiopexy, inguinal hernia repair, or tonsillectomy +/- adenoidectomy +/- ear tubes under general anesthesia.
* Primary language must be English, Spanish, Arabic, Nepali, or Somali.

Exclusion Criteria:

* ASA ≥ 3
* chronic pain condition
* inpatient
* regional anesthesia.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Caregivers of children age 3-17 presenting for surgery at NCH.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
sTOFHLA survey | From enrollment to prior to surgery start.
  Short Test of Functional Health Literacy in Adults
  Raw Score (0-36) Inadequate Functional Health Literacy (0-16) Marginal Functional Health Literacy (17-22) Adequate Functional Health Literacy (23-36)

SECONDARY OUTCOMES:
6-STAI | From enrollment to prior to surgery start.
  6-item State Trait Anxiety Inventory survey 6 question survey on 1-4 Likert Scale (Not at all, Somewhat, Moderately, Very Much) with total scores ranging from 6-24. Higher scores indicate greater anxiety.
Postoperative patient pain scores | Perioperative
  Pain Scores using Numeric Rating Scale (NRS) on a scale of 0-10; Visual Analog Scale (VAS) on a scale of 0 "No Pain" to 10 "Worst Pain"; Wong-Baker FACES Pain Rating Scale; FLACC Scale for non-verbal or pre-verbal patients. Higher scores indicate higher levels of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No